CLINICAL TRIAL: NCT04296175
Title: A Prospective, Single Center, Randomized, Open-labled Stage III Clinical Trial Comparing the Efficacy and Safety of Anthracyclin Followed by Weekly Paclitaxel Versus Dose-dense Anthracyclin Followed by Weekly Paclitaxel Versus Dose-dense Anthracyclin Followed by Weekly Paclitaxel Combined With Carboplatin for High-risk, Triple-negative Early Breast Cancer
Brief Title: Carboplatin Intensified Chemotherapy for TRIple NEgative Breast Cancer(CITRINE)
Acronym: CITRINE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1807187-2
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Triple-negative Breast Cancer
Keywords: dose-dense chemotherapy; Carboplatin; High-risk, Triple-negative Early Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Epirubicin; Paclitaxel; Carboplatin

STUDY DESIGN:
Intervention Model Description: 1:1 randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional group (Active Comparator): epirubincin 90mg/m2 d1 and CTX 600mg/m2 d1, every 2 or 3 weeks followed by paclitaxel 80mg/m2 d1,d8,d15, every 3 weeks.
  Interventions: Drug: Epirubicin; Drug: CTX; Drug: Paclitaxel
- carboplatin group (Experimental): epirubincin 90mg/m2 d1 and CTX 600mg/m2 d1, every 2 weeks followed by paclitaxel 80mg/m2 and carboplatin AUC=2 d1,d8,d15, every 4 weeks.
  Interventions: Drug: ddEpirubicin; Drug: ddCTX; Drug: Paclitaxel(with carbo); Drug: Carboplatin

INTERVENTIONS:
Drug: Epirubicin — 90mg/m2, d1 every 2 or 3 weeks
  Arms: conventional group
Drug: CTX — 600mg, d1 every 2 or 3 weeks
  Arms: conventional group
Drug: Paclitaxel — 80mg/m2,d1,d8,d15, every 3 weeks
  Arms: conventional group
Drug: ddEpirubicin — 90mg/m2, d1 every 2 weeks
  Arms: carboplatin group
Drug: ddCTX — 600mg, d1 every 2 weeks
  Arms: carboplatin group
Drug: Paclitaxel(with carbo) — 80mg/m2,d1,d8,d15, every 4 weeks
  Arms: carboplatin group
Drug: Carboplatin — AUC=2,d1,d8,d15, every 4 weeks
  Arms: carboplatin group

SUMMARY:
This is a prospective, single center, randomized, open-labled stage III clinical trial comparing the efficacy and safety of anthracyclin followed by weekly paclitaxel versus dose-dense anthracyclin followed by weekly paclitaxel versus dose-dense anthracyclin followed by weekly paclitaxel combined with carboplatin for high-risk, triple-negative early breast cancer.

DETAILED DESCRIPTION:
This is a prospective, single center, randomized, open-labled stage III clinical trial comparing the efficacy and safety of anthracyclin followed by weekly paclitaxel versus dose-dense anthracyclin followed by weekly paclitaxel versus dose-dense anthracyclin followed by weekly paclitaxel combined with carboplatin for high-risk, triple-negative early breast cancer.High risk is defined as positive lymph nodes or negative lymph nodes but ki-67 is not less than 50%. We aim to explore whether the addition of carboplatin can improve the disease-free survival of early high-risk triple-negative breast cancer. At the same time, the experimental group's anthracyclines must be given in a dose-dense manner, while anthracyclines in the control group are dose-dense or not.

ELIGIBILITY:
Inclusion Criteria:

1. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
2. Histologically documented TNBC after early breast cancer surgery (absence of HER2, ER, and PR expression)
3. Has adequate organ function meeting the following criteria: (1) adequate bone marrow function: hemoglobin ≥ 90 g/L (no blood transfusion within 14 days); absolute neutrophil count ≥ 1.5 x 109 /L; platelet count ≥ 75 * 109 /L; (2)adequate liver and kidney function: Alanine Aminotransferase (ALT) ≤ 3×upper limit of normal (ULN), Aspartate Aminotransferase (AST) ≤ 3×ULN, Total Bilirubin (TBIL)≤ 1.5×ULN, serum creatinine ≤ 1×ULN#and with endogenous creatinine clearance rate of >50 ml/min (Cockcroft-Gault formula).
4. Women aged 18-70 years old;
5. Lymph nodes positive or lymph nodes negative but with ki67 no less than 50%
6. Have the cognitive ability to understand the protocol and be willing to participate and to be followed up
7. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures as outlined for each specific treatment arm

Exclusion Criteria:

1. Has received neoadjuvant therapy (include chemotherapy, targeted therapy, radiotherapy or endocrine therapy;
2. Has bilateral breast cancer;
3. Has previous history of additional malignancy, with the exception of adequately treated basal cell carcinoma and cervical carcinoma in situ.
4. Has metastatic breast cancer
5. Is pregnant, is breast feeding women, or women of childbearing age who cannot practice effective contraceptives;
6. Patients participating in other clinical trials at the same time;
7. Has severe organ dysfunction (cardiopulmonary liver and kidney) insufficiency, left ventricular ejection fraction (LVEF) < 50% (cardiac ultrasound); severe cardio cerebral vascular disease within the 6 months previous of randomization (such as unstable angina, chronic heart failure, uncontrolled hypertension with blood pressure>150/90mmgh, myocardial infarction, or cerebral blood vessel); diabetic patients with poor blood glucose control; patients with severe hypertension;
8. Has known allergy to taxane
9. Has severe or uncontrolled infection;
10. Has a history of psychotropic substance abuse and were unable to abandon drug habits, or those with history of mental disorders;
11. the researchers judged patients to be unsuitable for the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 808 (Estimated)
Dates: Start 2020-03-05 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 3 year

SECONDARY OUTCOMES:
overall survival | 3 year
distant disease free survival | 3 year
recurrence free survival | 3 year
Disease free survival | 5 year
overall survival | 5 year
recurrence free survival | 5 year
distant disease free survival | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, Professor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Liu Y, Gong Y, Zhu XZ, Liu GY, Yu KD, Yang F, Chen L, He M, Hu Z, Chen CM, Cao AY, Li JJ, Hou YF, Di GH, Wu J, Jiang YZ, Fan L, Wang ZH, Shao ZM. Effect of adjuvant carboplatin intensified chemotherapy versus standard chemotherapy on survival in women with high risk, early stage, triple negative breast cancer (CITRINE): randomised, open label phase 3 trial. BMJ. 2025 Dec 23;391:e085457. doi: 10.1136/bmj-2025-085457. PMID 41436191